CLINICAL TRIAL: NCT06878573
Title: Description of the Changes of Ocular Perfusion in Patients with Age-related Maculopathy or Diabetic Macula Edema After Intravitreal Aflibercept Injection Treatment
Brief Title: Change in Ocular Perfusion After Intravitreal Anti-VEGF in Patients with Age-related Maculopathy or Diabetic Macula Edema
Status: Completed | Type: Observational
Sponsor: Augenabteilung Allgemeines Krankenhaus Linz (Other)
Responsible Party: Sponsor
Other Study IDs: LSFG-aflibercept-ARMandDME
Record Dates: First submitted 2025-03-06; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Age Related Macular Degeneration; Diabetic Macular Edema
Keywords: ocular perfusion; laser speckle flowgraphy; anti-VEGF
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Age-related macular degeneration: Patients with neovascular age-related macular degeneration, requiring Anti-VEGF
  Interventions: Drug: Intravitreal Aflibercept Injection; Device: Laser speckle flowgraphy
- Patients with diabetic macular edema: Patients with diabetic macular edema, requiring Anti-VEGF
  Interventions: Drug: Intravitreal Aflibercept Injection; Device: Laser speckle flowgraphy

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection — After instillation of topical anesthesia (0.4% oxybuprocaine hydrochloride and lidocain; own production), sterilization of the eyelid (Betaisodona solution 11% povidone-iodine, Mundipharma, Limburg, Germany), and instillation of 1.25% povidone-iodine drops, 2.0 mg/0.05 mL of aflibercept (Eylea) will be injected into the vitreous cavity through a standard pars plana approach (3.5 mm posterior to the limbus) under sterile conditions.
Device: Laser speckle flowgraphy — The RetFlow consists of a fundus camera equipped with a diode laser at a wavelength of 830 nm and a digital charge-coupled device camera (750 x 360 pixels). A total of 118 images are acquired at a rate of 30 frames per second over a 4-second measurement period. The main output parameter of LSFG, mean blur rate (MBR), is calculated from the pattern of speckle contrast produced by the interference of a laser scattered by blood cells moving in the ocular fundus. MBR was calculated for the total ONH area, defined by a ellipsoid region of interest (ROI). By using the on-board software, the MBR will be calculated in the large vessels within the ONH (ONH-MV, "mean MBR of vascular area") and the tissue area containing the microvasculature (ONH-MT, "mean MBR of tissue area")

SUMMARY:
This prospective study will include patients with neovascular age-related macular degeneration or diabetic macular edema, scheduled for intravitreal aflibercept. Ocular perfusion will be measured by Laser Speckle Flowgraphy (LSFG). The parameter Mean Blur Rate (MBR) reflects erythrocyte flow velocity and serves as an indirect marker of perfusion. MBR will be measured at the optic nerve head (ONH). The devices software can analyze MBR in areas of major retinal vessels (MV) and in microperfusion areas (MT) separately. Measurements will be conducted on the day of the planned intravitreal injection and one and four weeks post-injection.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years,
* patients scheduled for an intravitreal injections with Aflibercept for treatment of DME or AMD.

Exclusion Criteria:

* ocular surgery (including intravitreal injection) during the 3 months preceding the study
* Ametropia > 6 Dpt
* any relevant ophthalmic diseases/conditions that could interfere with LSFG measurements (e.g. glaucoma, optic nerve head drusen, tilted disc, etc.).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasian patients scheduled for intravitreal Aflibercept because of age related macular degeneration or diabetic macular edema
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Mean blur rate in retinal vessels (MV) | Baseline; Week 1; Week 4;
  With the onboard software, MBR can be calculated in the large vessels within the ONH (ONH-MV, "mean MBR of vascular area")

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Ophthalmology, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No